CLINICAL TRIAL: NCT06623877
Title: Using Renal Elastography Measurements for Evaluation of Glomerulonephritis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmes Essam Mohamed, Specialist of nephrology, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 6121820722
Record Dates: First submitted 2024-09-24; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Evaluation of Biopcy Proven Glomerulonephritis Patients by Renal Shear Wave Elastography
Keywords: elastography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: biopcy proven glomerulonephritis patients not started specific treatement (Experimental): agroup of Biopcy proven glomerulonephritis patients not started specific treatement will undergo for renal shear wave elastography
  Interventions: Diagnostic Test: renal shear wave elastography
- Group B : healthy persons (Experimental): A group of healthy persons will undergo for renal shear wave elastography
  Interventions: Diagnostic Test: renal shear wave elastography

INTERVENTIONS:
Diagnostic Test: renal shear wave elastography — Renal shear wave elastography is a non-invasive ultrasound elastography technique that allows measurements of tissue stiffness. It provides real-time measurements of shear wave velocity (SWV) generated with an acoustic impulse, thereby providing quantitative information about tissue elasticity. Harder tissues have been shown to have higher SWV .
  Renal shear wave elastography will be done to both groups

SUMMARY:
All participants will clinically evaluated by history taking, full physical examination including body weight and assessment of fluid status, and blood and urine samples for lab analysis (serum creatinine, urea, sodium, potassium, corrected calcium, phosphorous, estimated glomerular filtration rate(GFR) by Cokcroft equation ((140 - age ) x body weight by Kg/creatinine by µmol )complete urine analysis including microscopic examination of urine , 24 hours urinary protein , haemoglobin level .

All participants will undergo renal shear wave elastography measurements. Values will be obtained from the upper, middle, and lower zones of each kidney. A total of six shear wave elastography measurements will be collected to get mean elastography values (MEVs) of each participant.

DETAILED DESCRIPTION:
We will collect results of MEV plus blood and urine samples of each participant then data will undergo statistical analysis to compare between MEV of healthy persons and biopcy proven glomerulonephritis patients

ELIGIBILITY:
a-inclusion criteria :

* adult patients aged 18 years old or more
* patients diagnosed as glomerulonephritis ( biopcy proven ) and not started specific tratement in Assiut University Hospitals

  b. Exclusion criteria:
* patient with urinary tract obstruction
* patient who has GN and started corticosteroid and/or immunosuppressive drugs
* patient who has congenital anomalies in renal system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
comparisons between the shear wave elastography measurements in GN patients and healthy persons . | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine,Assiut universty,Egypy, Asyut, Asyut Governorate, Egypt